CLINICAL TRIAL: NCT01958398
Title: Brief Alcohol Interventions With Mobile Phone Applications for University Students: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/1126-31/1
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Problematic Alcohol Use
Keywords: Randomized Controlled Trial; Alcohol; Internet; Mobile phone; Screening; Brief intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Promillekoll (Experimental): Smartphone app monitoring alcohol use with feedback.
  Interventions: Behavioral: Promillekoll
- PartyPlanner (Experimental): Smartphone-adapted web based app for simulating an event with alcohol consumption in advance, real time monitoring alcohol use with feedback during the event and the possibility to compare these two.
  Interventions: Behavioral: PartyPlanner
- Control (No Intervention): Untreated control group

INTERVENTIONS:
Behavioral: Promillekoll — Smartphone app monitoring alcohol use with feedback.
  Arms: Promillekoll
Behavioral: PartyPlanner — Smartphone-adapted web based app for simulating an event with alcohol consumption in advance, real time monitoring alcohol use with feedback during the event and the possibility to compare these two.
  Arms: PartyPlanner

SUMMARY:
Objectives: This study evaluates the efficacy of two mobile phone applications, Promillekoll and PartyPlanner among university government members at two universities in Stockholm, Sweden. The design is a three-armed randomized controlled design, and outcomes are measured in terms of changes in problematic alcohol use at follow up 7 weeks after study initiation and baseline data gathering. Both the Promillekoll and PartyPlanner apps feature real time registration of alcohol consumption and giving feedback of estimated blood alcohol concentration levels. Both apps inform and warn the user when the estimated alcohol level is above 0.6%, a level set that is below risky consumption levels. PartyPlanner additionally provides the possibility of simulating and planning an alcohol consumption event in advance and later on comparing it with the real time registration at the event.

Method: Participants with problematic alcohol use (AUDIT >7 for men and >5 for women) are randomized into one of three groups: 1. Access to Promillekoll, 2. Access to PartyPlanner and 3. Control group. Outcomes on alcohol use as well as information on the users' satisfaction with the app assigned to them gathered after 7 weeks.

The hypotheses are: 1. The groups receiving the Promillekoll and PartyPlanner interventions will reduce their alcohol use to a larger extent than the control group at follow-up compared to the baseline level. 2. The addition of the possibility to plan events beforehand (PartyPlanner) will lead to an increased decrease in alcohol consumption to only real-time use (Promillekoll).

DETAILED DESCRIPTION:
Background Brief interventions via the internet have been shown to reduce university students' alcohol intake. This study tested two smartphone applications (apps) targeting drinking choices on party occasions, with the goal of reducing problematic alcohol intake among Swedish university students.

Methods Students were recruited via e-mails sent to student union members at two universities. Those who gave informed consent, had a smartphone, and showed risky alcohol consumption according to the Alcohol Use Disorders Identification Test (AUDIT) were randomized into three groups. Group 1 had access to the Swedish government alcohol monopoly's app, Promillekoll, offering real-time estimated blood alcohol concentration (eBAC) calculation; Group 2 had access to a web-based app, PartyPlanner, developed by the research group, offering real-time eBAC calculation with planning and follow-up functions; and Group 3 participants were controls. Follow-up was conducted at 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Access to a smartphone running iOS or Android OS.
* AUDIT >7 for men or AUDIT >5 for women.

Exclusion Criteria:

* AUDIT <8 (men) or <6 (women)
* No access to a smartphone running iOS or Android OS.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4408 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in estimated Blood Alcohol Concentration (eBAC) | 7 weeks
  Change in Blood Alcohol Concentration estimated using Widmark's formula for Blood Alcohol Concentration estimation.

SECONDARY OUTCOMES:
AUDIT-C | 7 weeks
  The change in score for the first three AUDIT questions, as a measure of alcohol consumption only, referred to as the AUDIT-C.
Alcohol Use Disorders Identification Test (AUDIT) | 7 weeks
  Change in total AUDIT score, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems).

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neuroscience, Stockholm, Sweden

REFERENCES:
- [Result] Gajecki M, Berman AH, Sinadinovic K, Rosendahl I, Andersson C. Mobile phone brief intervention applications for risky alcohol use among university students: a randomized controlled study. Addict Sci Clin Pract. 2014 Jul 2;9(1):11. doi: 10.1186/1940-0640-9-11. PMID 24985342